CLINICAL TRIAL: NCT04373902
Title: Physiological-based Cord Clamping Versus Immediate Cord Clamping for Infants Born With Congenital Diaphragmatic Hernia: a Multicentre, Randomised Controlled Trial
Brief Title: Physiological-based Cord Clamping in Congenital Diaphragmatic Hernia
Acronym: PinC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Philip L.J. DeKoninck, Principal Investigator, Dr., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PinC CDH trial; NL7853 (Registry Identifier: NTR)
Record Dates: First submitted 2020-04-14; First posted 2020-05-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hernias, Diaphragmatic, Congenital; Hernia; Diaphragm Defect, Congenital; Pulmonary Hypertension
Keywords: Congenital diaphragmatic hernia; Perinatal stabilisation; Resuscitation; Pulmonary hypertension; Birth defect; Physiological-based cord clamping
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Hernia, Diaphragmatic; Hypertension, Pulmonary; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physiological-based cord clamping (Experimental): In PBCC, the Concord will be placed next to the bed of the mother and all equipment will be checked before the second stage of labour has started. The infant will be placed on the platform of the Concord immediately after birth, avoiding any traction or pressure on the cord and avoiding heat loss by radiation heating. The umbilical cord will not be clamped until the infant is considered respiratory stable, which is defined as the presence of a heart rate >100 bpm and preductal oxygen saturation >85%, while using an fraction of inspired oxygen (FiO2) of <0.5. The minimum and maximum times of cord clamping are three and ten minutes after birth, respectively. Oxytocin administration will be postponed until after cord clamping if there are no obstetric concerns. At any time, the attending neonatologist and obstetrician can decide that PBCC should not be performed or be interrupted. In that case, the infant can be placed on the standard resuscitation table for (further) stabilisation.
  Interventions: Procedure: Physiological-based cord clamping
- Immediate cord clamping (No Intervention): In the immediate cord clamping group, the cord will be clamped immediately after birth. The infant will then be transferred to the standard neonatal resuscitation table. After cord clamping, all infants will be managed according to the standardised neonatal management protocol for infants with a CDH, which is a consensus of current clinical guidelines by the CDH EURO consortium.

INTERVENTIONS:
Procedure: Physiological-based cord clamping — See 'Arm'
  Arms: Physiological-based cord clamping

SUMMARY:
Pulmonary hypertension is a major determinant of postnatal survival in infants with a congenital diaphragmatic hernia (CDH). The current care during the perinatal stabilisation period in infants born with this rare birth defect might contribute to the development of pulmonary hypertension after birth - in particular umbilical cord clamping before lung aeration. An ovine model of diaphragmatic hernia demonstrated that cord clamping after lung aeration, called physiological-based cord clamping (PBCC), avoided the initial high pressures in the lung vasculature while maintaining adequate blood flow, thereby avoiding vascular remodelling and aggravation of pulmonary hypertension. The investigators aim to investigate if the implementation of PBCC in the perinatal stabilisation period of infants born with a CDH could reduce the incidence of pulmonary hypertension in the first 24 hours after birth.

The investigators will perform a multicentre, randomised controlled trial in infants with an isolated CDH. Before birth, infants will be randomised to either PBCC or immediate cord clamping, stratified by treatment centre and severity of pulmonary hypoplasia on antenatal ultrasound. For performing PBCC a purpose-designed resuscitation module (the Concord Birth Trolley) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Left-sided CDH
* Isolated CDH: no associated structural or genetic abnormalities that are diagnosed before birth
* Gestational age at delivery ≥35.0 weeks
* Parental written informed consent

Exclusion Criteria:

* Right-sided or bilateral CDH
* Gestational age at delivery <35.0 weeks
* Maternal contraindications: anterior placenta praevia, placental abruption
* High urgency caesarean section, with intended interval to delivery <15 min
* Cases that have been treated during pregnancy with experimental drug therapy aiming to decrease the occurrence of pulmonary hypertension
* Twin pregnancies in which the infant diagnosed with a CDH is born first
* Multiple birth >2 (triplets or higher order)

Min Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with pulmonary hypertension diagnosed in the first 24 hours after birth. | First 24 hours after birth
  Pulmonary hypertension is present if at least 2 of the following 4 criteria are present or if the infant requires extracorporeal membrane oxygenation (ECMO) in the first 24 hours after birth:
  1. Right ventricular systolic pressure (RVSP) ≥2/3 systemic systolic pressure*
  2. Right ventricle (RV) dilatation/septal displacement or RV dysfunction +/- left ventricle (LV) dysfunction*
  3. Pre-post ductal SpO2 difference >10% for at least 15 consecutive minutes
  4. Oxygenation Index >20** *as found on first ultrasound in first 24 hours after birth; **highest value measured in first 24 hours after birth
  The following echocardiographic parameters will be collected to objectify these criteria:
  * RV size
  * Pulmonary artery acceleration time (PAAT), right ventricular ejection time (RVET), PAAT:RVET ratio
  * Intraventricular septum configuration
  * LV systolic eccentricity index
  * Mean airway pressure
  * PaO2
  * FiO2
  * Preductal+postductal SpO2

SECONDARY OUTCOMES:
Neonatal: mortality before discharge from the tertiary care hospital | From birth till discharge from the tertiary care hospital, through study completion an average of one year
  Number of patients that died before discharge
Neonatal: presence of 3 or more criteria for pulmonary hypertension or extracorporeal membrane oxygenation within 24 hours after birth | The first 24 hours after delivery
  Number of patients with 3 or more criteria or ECMO
Neonatal: number of patients requiring ECMO therapy | From admission to the ICU until the date of death or the date of discharge home, whichever came first
  Number of patients requiring ECMO therapy
Neonatal: number of days of duration of supplemental oxygen need | From admission to the ICU until the date of discharge to another ward or home, whichever came first,through study completion an average of one year
  Number of days of duration of supplemental oxygen need
Neonatal: number of days of duration of mechanical ventilation | From admission to the ICU until the date of discharge to another ward or home, whichever came first,through study completion an average of one year
  Number of days of duration of mechanical ventilation
Neonatal: duration of admission to the tertiary care hospital | From admission to the ICU until the date of discharge to another ward or home, whichever came first
  Number of days of admission to the tertiary care hospital
Maternal: number of patients with postpartum haemorrhage | The first 24 hours after delivery
  Postpartum haemorrhage is defined as estimated blood loss >1000 mL

CONTACTS AND LOCATIONS:
Locations (9):
- Monash University, Melbourne, Australia
- Medical University Graz, Graz, Austria
- University Hospitals leuven, Leuven, Belgium
- Germany (2):
  - Universitätskrankenhaus Bonn, Bonn
  - Universitätsklinik Mannheim, Mannheim
- Ospedale Pediatrico Bambino Gesu, Rome, Italy
- Netherlands (2):
  - Radboudumc University Medical Center, Nijmegen
  - Erasmus MC University Medical Center - Sophia Children's Hospital, Rotterdam
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horn-Oudshoorn EJJ, Vermeulen MJ, Knol R, Bout-Rebel R, Te Pas AB, Hooper SB, Otter SCMC, Wijnen RMH, Crossley KJ, Rafat N, Schaible T, de Boode WP, Debeer A, Urlesberger B, Roberts CT, Kipfmueller F, Capolupo I, Burgos CM, Hansen BE, Reiss IKM, DeKoninck PLJ. Multicentre, randomised controlled trial of physiological-based cord clamping versus immediate cord clamping in infants with a congenital diaphragmatic hernia (PinC): statistical analysis plan. Trials. 2024 Mar 20;25(1):198. doi: 10.1186/s13063-024-08027-7. PMID 38509614
- [Derived] Horn-Oudshoorn EJJ, Knol R, Vermeulen MJ, Te Pas AB, Hooper SB, Cochius-den Otter SCM, Wijnen RMH, Crossley KJ, Rafat N, Schaible T, de Boode WP, Debeer A, Urlesberger B, Roberts CT, Kipfmueller F, Reiss IKM, DeKoninck PLJ. Physiological-based cord clamping versus immediate cord clamping for infants born with a congenital diaphragmatic hernia (PinC): study protocol for a multicentre, randomised controlled trial. BMJ Open. 2022 Mar 18;12(3):e054808. doi: 10.1136/bmjopen-2021-054808. PMID 35304395